CLINICAL TRIAL: NCT01730131
Title: Natural History Study of Progressive Multifocal Leukoencephalopathy (PML)
Status: Recruiting | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130017; 13-N-0017
Record Dates: First submitted 2012-11-17; First posted 2012-11-21 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01-26

CONDITIONS: Progressive Multifocal Leukoencephalopathy
Keywords: Encephalitis; Immune Reconstitution Syndrome; Human Immunodeficiency Virus; Multiple Sclerosis; Natural History
MeSH Terms: conditions — Leukoencephalopathy, Progressive Multifocal; Encephalitis; Immune Reconstitution Inflammatory Syndrome; Acquired Immunodeficiency Syndrome; Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Patients at Risk for PML: Participants with impaired immune function from any cause and considered at risk for PML
- Healthy Volunteers: Healthy volunteers without impaired immune function
- PML Patients: Participants with PML

SUMMARY:
Background:

- Progressive multifocal leukoencephalopathy (PML) is a severe viral infection of the brain. It is caused by JC virus. Many people have this virus in their bodies all their life, but it is usually kept in check by their immune system. If the immune system does not work right because of a disease or medication, the virus becomes active and can damage cells in the brain. Not much is known about PML or how it affects the immune system. Researchers want to study people with PML to better understand the natural history of the disease.

Objectives:

- To study the natural history of PML.

Eligibility:

- Individuals at least 2 years of age who have PML.

Design:

* Participants will be screened with a physical exam, medical history, and imaging studies.
* Participants will have several visits to the National Institutes of Health Clinical Center. There will be an initial visit, monthly visits for the next 6 months, a 12-month visit, and possible visits afterward.
* At the initial visit, participants will give blood, urine, and spinal fluid samples. They will also have neurological tests and imaging studies of the brain.
* For the next five visits, participants will give blood and urine samples. They will also have neurological tests and imaging studies of the brain.
* The 6-month and 12-month visits will repeat the tests from the initial visit.
* Other optional procedures include bone marrow samples and skin biopsies. Additional blood tests and imaging studies may be performed.
* Treatment will not be provided as part of this study.

DETAILED DESCRIPTION:
The objective of this study is to examine the risk factors and natural course of JCV infection and progressive multifocal leukoencephalopathy (PML). PML is a devastating, demyelinating neurological disease affecting the brain of patients with a compromised immune system. It is caused by reactivation of JC virus (JCV), a small DNA virus that infects the majority of the population without clinical significance. There are currently no treatments available for PML.

We plan to study patients with suspected or confirmed PML with different underlying conditions including patients on immune-modulatory therapies for multiple sclerosis (MS), rheumatologic diseases or other autoimmune diseases, as well as patients with HIV infection or other conditions leading to a compromised immune system. Patients will be seen at defined time points during their disease course and detailed assessments will be performed to collect clinical and imaging data. Blood, cerebrospinal fluid (CSF) and urine will also be collected at these time points to evaluate the behavior and biology of the JCV and the patients immune responses to the infection. These tests will lead to a better understanding of the pathophysiology of PML and the course of this disease in different patient groups. Additionally, we will recruit a patient control cohort represented by patients with impaired immune function for any cause and considered at risk for development of PML, and a healthy volunteer cohort. The purpose of these additional cohorts is to explore and validate biomarkers for risk of development of PML and early diagnosis. Additionally, the healthy volunteer cohort may be screened and evaluated as possible donors of peripheral blood mononuclear cells (PBMC) for manufacture of virus-specific T cells.

The detailed characterization described above will be used to help identify:

1. Clinical, imaging, and/or laboratory features pathognomonic of JCV infection and disease course that may aid in earlier diagnosis and appropriate intervention
2. Clinical, imaging, and/or laboratory features of JCV infection and disease course that are predictive of clinical outcomes

This information will be integrated to develop a clinically relevant, disease-specific assessment scale of PML, which is currently not available. Such a scale would be a useful tool for the clinical management of patients (i.e., for development of standards of care), as well as for clinical trial design and interpretation.

The long-term objectives of this study are to improve the understanding of the disease course and underlying pathophysiology, to identify subgroups with different prognosis and/or susceptibility to interventions, and to help identify therapeutic targets and/or intervention strategies. Equally important, these efforts will allow development of a repository of cryopreserved biological samples that will be used for validation of candidate biomarkers in future studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Suspected or confirmed PML
  2. MRI compatible with PML
  3. Able to participate in the studies and follow-up required by the protocol
  4. At least 2 years old

EXCLUSION CRITERIA:

1. Significant condition, which in the judgment of the principal investigator, would make participation in the diagnostic and research parts of evaluation impossible or risky
2. Medical contraindication to MRI (i.e., devices such as a cardiac pacemaker or infusion pump, other metallic implants, metallic foreign objects, body piercings that cannot be removed)
3. Pregnancy
4. Inability to provide informed consent, either directly or via legally authorized representative (LAR)
5. Unwillingness to consent for collection of biological samples or their cryopreservation

Ages: 2 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary clinical for participants that have PML or at risk for PML and community sample/healthy relatives for healthy volunteers.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2012-11-08 (Actual); Primary Completion 2052-01-01 (Estimated)

PRIMARY OUTCOMES:
To characterize the baseline presentation of patients with JCV infection and/or PML with regard to clinical, radiological, immunological, genetic and viral features. | one year following last enrollment
  1. Characterization of distinctive imaging features to differentiate between actively progressing PML, PML-IRIS/inflammatory PML and inactive PML2. Characterization of distinctive clinical features to differentiate between actively progressing PML, PML-IRIS/inflammatory PML, and inactive PML3. Characterization of immune and virological features to differentiate between actively progressing PML, PML-IRIS/inflammatory PML, and inactive PML4. Characterization of immune and virological differences across PML patient populations with different underlying disease, subjects at risk for developing PML, and healthy individuals5. Characterization of genetic susceptibility for development of PML

SECONDARY OUTCOMES:
To longitudinally follow patients with JCV infection and/or PML with thorough characterization of their clinical course, imaging correlates, immunological markers, and viral studies | one year following last enrollment
  1. Temporal correlation between clinical course and imaging and/or laboratory measures2. To identify biomarkers that can predict long-term outcome and response to treatment interventions3. To develop a clinically relevant assessment scale for PML that identifies milestones of disease progression4. To develop a repository of cryopreserved biological samples that will be used for validation of candidate biomarkers in future studies5. To characterize the immune profile in blood and CSF of patients with PML6. To determine the eligibility of PML patients for participation in other studies7. To screen and evaluate healthy subjects as donors for manufacture of virus-specific T cells (to be administered to patients under separate, dedicated protocol)

CONTACTS AND LOCATIONS:
Overall Officials: Irene CM Cortese, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Cinque P, Koralnik IJ, Gerevini S, Miro JM, Price RW. Progressive multifocal leukoencephalopathy in HIV-1 infection. Lancet Infect Dis. 2009 Oct;9(10):625-36. doi: 10.1016/S1473-3099(09)70226-9. PMID 19778765
- [Background] Padgett BL, Walker DL, ZuRhein GM, Eckroade RJ, Dessel BH. Cultivation of papova-like virus from human brain with progressive multifocal leucoencephalopathy. Lancet. 1971 Jun 19;1(7712):1257-60. doi: 10.1016/s0140-6736(71)91777-6. No abstract available. PMID 4104715
- [Background] Gheuens S, Pierone G, Peeters P, Koralnik IJ. Progressive multifocal leukoencephalopathy in individuals with minimal or occult immunosuppression. J Neurol Neurosurg Psychiatry. 2010 Mar;81(3):247-54. doi: 10.1136/jnnp.2009.187666. Epub 2009 Oct 14. PMID 19828476
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-N-0017.html